CLINICAL TRIAL: NCT04454034
Title: Arthroscopic Synovectomy Combined With DMARDs in the Treatment of Refractory Elbow Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019072
Record Dates: First submitted 2020-06-27; First posted 2020-07-01 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2020-06

CONDITIONS: Rheumatoid Arthritis of Ankle
Keywords: Rheumatoid Arthritis; Arthroscopic Synovectomy
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Group1: The refractory elbow RA who undergo arthroscopic synovectomy
  Interventions: Procedure: arthroscopic synovectomy

INTERVENTIONS:
Procedure: arthroscopic synovectomy — arthroscopic synovectomy

SUMMARY:
Rheumatoid arthritis (RA) is an autoimmune disease characterized by chronic and aggressive polyarthritis. The prevalence of RA in China is about 0.42%. Arthroscopic synovectomy (AS) is an important method to save the function of joint in the treatment of refractory RA. The clinical trial is to study the value of AS combine with DMARDs in the early stage of refractory RA.

ELIGIBILITY:
Inclusion Criteria:

* The patients who fulfilled the 1987 ACR（American College of Rheumatology) or 2010 ACR/EULAR（European League Against Rheumatism） RA classification criteria.
* The age is more than 18 years old and less than 60 years old.
* They received stable traditional DMARDs (including Chrysopidae, leflunomide, sulfasalazine, hydroxychloroquine, eilamod) or biological dmrads (including tumor necrosis factor antagonists, IL(Interleukin)-6 receptor antagonists, CD20 monoclonal antibodies) for at least 6 months.
* The disease is still in the active stage, which means the disease activity score (DAS28) is more than 3.2, and the elbow joint function is obviously limited.
* The patient agreed to undergo arthroscopic synovectomy.
* No contraindications were found.

Exclusion Criteria:

* The disease is in remission.
* The patient has contraindications.
* Arthroscopic synovectomy was performed in different patients.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: the patients who fullfill the Eligibility Criteria
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
ACR70 remission | 6 months after surgery
  the percent of patients who meet ACR70 remission

SECONDARY OUTCOMES:
Disease Activity Score (DAS) 28-erythrocyte sedimentation rate (ESR) (range 0-9.4) | 1,3,6 and 12 months after surgery
  Remission: 2.6 Low activity: 2.6 to ,3.2 Moderate activity: 3.2 to 5.1 High activity: .5.1
tender joint count | 1,3,6 and 12 months after surgery
  the number of tender joints
swollen joint count | 1,3,6 and 12 months after surgery
  the number of swollen joints

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Univerisity Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided